CLINICAL TRIAL: NCT04585360
Title: Psychiatric Manifestations Associated With Behcet's Disease
Acronym: PSYCHO-B7
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-A01819-48
Record Dates: First submitted 2020-10-09; First posted 2020-10-14 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Behçet's Disease; Psychiatric Disorders
Keywords: NeuroBehçet; Anxiety; Depression; Tiredness
MeSH Terms: conditions — Behcet Syndrome; Mental Disorders; Anxiety Disorders; Depression; Fatigue | interventions — Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with Behcet disease: adult patient with Behcet's disease followed regularly in the internal medicine department of Bicetre
  Interventions: Other: Questionnaires evaluating anxiety and depression symptoms, tiredness, and quality of life

INTERVENTIONS:
Other: Questionnaires evaluating anxiety and depression symptoms, tiredness, and quality of life — Realization of specific questionnaires evaluating:
  * psychiatric symptoms (self-assessment according to the SLC-90R questionnaire and hetero-assessment by the internist doctor of the center according to the M.I.N.I. questionnaire)
  * fatigue (Multidimensional Fatigue Inventory (MFI-20), French version, in self-assessment)
  * quality of life (SF36 self-assessment questionnaire)

SUMMARY:
The psychoBehçet'study is aimed at evaluating the psychological and neurocognitive symptoms in 25 consecutive patients followed for Behçet's disease. This is a monocentric, observational, non interventional study.

DETAILED DESCRIPTION:
Patients will be evaluated during a day-care facility for Behçet's disease activity together with evaluation of anxiety and depression symptoms (SCL90-R and MINI assessments), fatigue (MFI) and quality of life (SF36).

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female
* Regular follow-up in the internal medicine department of Bicetre hospital
* Diagnosed with Behçet's disease

Exclusion Criteria:

* Refusal to participate in the study
* Poor command of the French language
* Patients under legal protection
* Pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient regularly monitored in the internal medicine department of Bicêtre
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
SCL90-R questionnaire | Inclusion visit
  Anxiety/depression symptoms questionnaire

SECONDARY OUTCOMES:
MINI questionnaire | Inclusion visit
  Anxiety/depression symptoms questionnaire
Multidimensional Fatigue Inventory (MFI-20) questionnaire | Inclusion visit
  Tiredness assessment
SF36 questionnaire | Inclusion visit
  Quality of life
BSAS/BDCAF evaluation | Inclusion visit
  Behçet's disease activity

CONTACTS AND LOCATIONS:
Overall Officials: NOEL NN Nicolas, MD PhD, Principal Investigator — APHP, Hôpital Bicetre
Locations (1):
- Internal medecine department, Le Kremlin-Bicêtre, Val de Marne, France

IPD SHARING:
Plan to Share IPD: No